CLINICAL TRIAL: NCT06059014
Title: A Multicentric, Single Arm, Open-label, Phase I/II Study Evaluating PSMA Targeted Radionuclide Therapy in Adult Patients with Metastatic Clear Cell Renal Cancer
Brief Title: Phase I/II Study Evaluating PSMA Targeted Radionuclide Therapy in Adult Patients with Metastatic Clear Cell Renal Cancer
Acronym: PRadR
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study not feasible, patient accrual rate too low
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET22-313
Record Dates: First submitted 2023-09-18; First posted 2023-09-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Radiopharmaceuticals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-PSMA-1 (Experimental): Radiopharmaceutical - injectable solution
  Interventions: Drug: 177Lu-PSMA-1 (radiopharmaceutical)

INTERVENTIONS:
Drug: 177Lu-PSMA-1 (radiopharmaceutical) — 7.4 GBq (or 5.9 GBq in case of lower actvity) of 177Lu-PSMA-1, every 6 weeks for 4 administirations

SUMMARY:
This study is an open label Phase I/II study conducted according to a Fleming design, investigating the safety and the efficacy of 4 IV injections of 177Lu-PSMA-1 in patients with metastatic clear cell renal cancer.

This trial is divided in 2 parts:

* A safety run-in part aiming to assess the safety of 177Lu-PSMA-1 (with 6 patients treated at the starting activity = 7.4 GBq of 177Lu-PSMA-1, every 6 weeks (Q6W) for 4 administrations). If more than one patient experiences a ST during the first cycle of therapy (6 weeks), then a lower activity of 177Lu-PSMA-1 will be evaluated in an additional cohort of 6 patients (5.9 GBq). The 6 patients from this safety run-in step, treated at the activity selected for phase II, will be included in the evaluation of Phase II part.
* A Phase II part aiming to assess the clinical activity of 177Lu-PSMA-1

DETAILED DESCRIPTION:
Despite the improvement in the management of metastatic clear-cell renal cell carcinoma (mccRCC) with antiangiogenic agent and immunotherapy, there is still an unmet need for patients who progress under these therapies. Indeed, there is currently no standard treatment for patients beyond the 2nd line of treatment in the advanced/metastatic setting. Prostate Specific Membrane Antigen (PSMA) is highly expressed in neovessels of various solid tumors including RCC: 86% of ccRCC.Higher grade and stage, metastatic and lethal ccRCC showed higher PSMA expression in tumor vessels, reflecting tumor prognosis. PSMA may be a target expressed in metastatic ccRCC for radionuclide therapy using PSMA Ligands Radiolabeled with Lutetium-177 (PRLT). 177Lu-PSMA delivers ß-particle radiation to PSMA-expressing cells and the surrounding microenvironment with demonstrated efficacy in metastatic prostate cancer. In multitreated prostate cancer patients, the additional effect of 177Lu-PSMA-617 compared to best standard of care alone led to a 4-month OS benefit, with an estimated 38% reduction in risk of death in the 177Lu-PSMA-617 arm compared to the best standard of care arm (median OS 15.3 months versus 11.3 months respectively, hazard ratio [HR]: 0.62, p<0.001).

A phase I/II study will be conducted to evaluate the tolerability and efficacy of 177Lu-PSMA-1 in patients presenting with a PSMA-positive mccRCC selected through 68Ga-PSMA PET. Only patients with tumor tracer uptake greater than background will be treated with 4 cycles of 7.4 GBq of 177Lu-PSMA-1 every 6 weeks.

This study is an open label Phase I/II study conducted according to a Fleming design, investigating the safety and the efficacy of 177Lu-PSMA-1 repeated cycles in patients with metastatic ccRCC.

The study is divided in 2 parts:

• A safety run-in part aiming to assess the safety of 177Lu-PSMA-1: The study will begin with a safety run-in of 6 patients treated with 7.4 GBq of 177Lu-PSMA1 [starting activity], IV, q6W for 4 administrations.

If more than one patient experiences severe toxicity during the first cycle, then a lower activity of 177Lu-PSMA-1 will be evaluated in an additional cohort of 6 patients (5.9 GBq).

The 6 patients enrolled in this safety run-in step treated at the selected activity for phase II will be included in the evaluation of Phase II part.

• A Phase II part aiming to assess the clinical activity of 177Lu-PSMA-1

Patients will be treated and followed-up as following :

Selection step -68Ga-PSMA PET:

A selection step is mandatory for all patients in order to evaluate the PSMA expression in tumor lesions through 68Ga-PSMA PET and according to local imaging review. Only patients with PSMA expressing tumors will be eligible to the treatment step according eligbility

Treatment step:

Eligible patients will be treated with 177Lu-PSMA-1 (initial activity: 7.4 GBq), intravenously (IV) for 4 administrations every 6 weeks.

Assessment step:

To assess tumor response according to RECIST V1.1, imaging will be performed at baseline, at W9, at W24, then every 12 weeks up to 1 year after the first administration and then every 24 weeks until progression, death, loss to follow-up, or overall study completion, whichever is earliest. Survival status will be documented for all patients until death or overall study completion at least 12 months after the last patient.

ELIGIBILITY:
Inclusion Criteria:

I1. Male or female patients aged ≥ 18 years at time of informed consent signature.

I2. Patient with histologically confirmed diagnosis of metastatic clear cell renal cell carcinoma (mccRCC) previously treated by at least 2 lines of therapy in the advanced/metastatic setting including at least 1 line of anti-VEGFR and 1 line of immunotherapy.

I3. Patient with documented radiological disease progression at the time of inclusion with measurable disease as per RECIST v1.1.

I4. Patient with PSMA-PET positive lesions (68Ga-PSMA-PET):

* For patient with only extrahepatic disease: ≥ 50% of positive extrahepatic metastatic lesions
* For patient with both extra-hepatic and liver metastasis: ≥ 50% of positive extrahepatic metastatic lesions and ≥ 80 % of positive supracentimetric liver metastatic lesions.
* For patient with only liver metastatic lesions: ≥ 80 % of positive supracentimetric lesions.

I5. Life expectancy ≥ 3 months.

I6. Eastern Cooperative Oncology Group performance status 0, 1 or 2.

I7. Demonstrate adequate organ function as defined in the protocol.

I8. Women of child-bearing potential must have a negative urine pregnancy test at screening (within 72 hours prior C1D1) and must agree to use 1 effective form of contraception from the time of the treatment period and of the negative pregnancy test up to 6 months after the last administration of study drug. Effective forms of contraception are listed in the protocol.

I9. Fertile males must use highly effective contraception during the dosing period and through 6 months after final administration of study drug.

I10. Patient should be able and willing to comply with study visits and procedures as per protocol.

I11. Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.

I12. Patients must be covered by medical insurance.

Exclusion Criteria:

E1. Patients with known active central nervous system (CNS) metastases and/or epidural metastases. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to C1D1 and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids (at doses higher than 10 mg/d of methylprednisolone or equivalent) for at least 4 weeks prior to C1D1.

E2. Patients previously treated with any radiopharmaceutical, excluding 68Ga-PSMA required during screening for this protocol.

E3. Persisting toxicities related to previous anti-cancer therapy which were not resolved to grade ≤1 (except: anaemia provided that criterion I7 is met) and /or any persistent irAE of any grade (except adequately controlled irAE (e.g: with replacement therapy for endocrine irAE)).

E4. History, within 2 years, of cancer other than renal cancer, except for basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, localized prostate cancer.

E5. History of idiopathic pulmonary fibrosis, non-infectious pneumonitis, interstitial lung disease that required steroids or has current pneumonitis, interstitial lung disease, drug-induced pneumonitis, or evidence of active pneumonitis on screening chest CT scan.

E6. Prior therapy or a need to be treated with a forbidden concomitant/concurrent therapies/procedure as defined per protocol.

E7. Patients with clinically significant hematuria, hematemesis, or hemoptysis exceeding 0.5 teaspoon (2.5 mL) of red blood, as well as those with a history of coagulopathy or other significant bleeding (e.g., pulmonary hemorrhage) within the 3 months prior to the initiation of the study treatment. Patients receiving anticoagulation medication will be eligible only if the dosage and route of administration have remained stable since at least 2 weeks prior to C1D1.

E8. Patients with an active uncontrolled infection. E9. Women pregnant or breastfeeding. E10. Patients placed under a legal protection regimen such as: Judicial Safeguards, curatorship or guardianship

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Severe Toxicities (ST) (for Phase1 part) | during the first 6 weeks of treatment
  Incidence of Severe Toxicities (ST) defined as specific adverse events (AEs) graded using NCI-CTCAE V5.0 occurring during the ST period (i.e. the 6 first weeks) and assessed as related to study drug and considered clinically significant. The sepcific adverse events are defined in the protocol.
Disease Control Rate after 24 weeks of treatment (DCR24w) (for Phase II part) | at 24 weeks of treatment
  Disease Control Rate after 24 weeks of treatment (DCR24w) is defined as the rate of patients with a stable disease, a complete or partial response according to RECIST v1.1.after 24 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Leon Berard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kryza D, Vinceneux A, Bidaux AS, Garin G, Tatu D, Cropet C, Badel JN, Perol D, Giraudet AL. A multicentric, single arm, open-label, phase I/II study evaluating PSMA targeted radionuclide therapy in adult patients with metastatic clear cell renal cancer (PRadR). BMC Cancer. 2024 Feb 1;24(1):163. doi: 10.1186/s12885-023-11702-8. PMID 38302933